CLINICAL TRIAL: NCT00598988
Title: Acupuncture for Infectious Mononucleosis Trial
Acronym: AIM
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Difficulty with recruitment
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6866
Record Dates: First submitted 2007-12-04; First posted 2008-01-23 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2017-05

CONDITIONS: Infectious Mononucleosis
Keywords: infectious mononucleosis, mono, acupuncture
MeSH Terms: conditions — Infectious Mononucleosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): Traditional Chinese acupuncture in conjunction with standard medical care
  Interventions: Procedure: traditional Chinese acupuncture
- Standard medical care (Active Comparator): standard medical care
  Interventions: Other: standard medical care

INTERVENTIONS:
Procedure: traditional Chinese acupuncture — 10 treatments over 6 weeks
  Arms: Acupuncture
Other: standard medical care — standard care as provided by primary physician
  Arms: Standard medical care

SUMMARY:
The purpose of this study is to investigate feasibility issues related to conducting an acupuncture study in a population of adolescents and young adults with infectious mononucleosis. Additionally, this study will provide preliminary data regarding treatment parameters (acupuncture and standard care) and outcomes (i.e. fatigue).

DETAILED DESCRIPTION:
This study examines the feasibility of treating adolescents and young adults diagnosed with infectious mononucleosis with acupuncture. Additionally, this study will provide preliminary data regarding treatment parameters (acupuncture and standard care) and outcomes (i.e. fatigue).

ELIGIBILITY:
Inclusion Criteria:

* mono diagnosis confirmed by lab test
* 21 days or less between start of symptoms and diagnostic test
* presence of fatigue of at least 4/11 (by Chalder Fatigue Questionnaire)
* no other illnesses present
* meets residency requirement

Exclusion Criteria:

* insufficient communication in English
* unable to begin acupuncture within 21 days of diagnostic test
* acupuncture use currently or in the preceding 3 months
* currently under the care of a TCM practitioner
* unwilling to be randomized

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Chalder Fatigue Questionnaire | 12 weeks

SECONDARY OUTCOMES:
MOS SF-36 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Vohra, MD, MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided